CLINICAL TRIAL: NCT03950999
Title: Pain and Placebo - a Study to Examine Relations Between Pain Reporting Accuracy and the Response to Experimental Placebo Model
Brief Title: Experimental Pain Reporting Accuracy and Placebo Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Roi Treister, Head of The Clinical Pain Innovation Lab, University of Haifa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 273/17
Record Dates: First submitted 2019-05-07; First posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Healthy; Placebo Effect; Pain
Keywords: Focus analgesia selection test (FAST); Placebo effect; Experimental pain variability
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): Each subject underwent baseline assessment of pain reporting accuracy (FAST). Thereafter, the placebo response was assessed using tonic heat stimuli delivered at fixed temperature of 44, 46.5, and 48°C which evoke mild, moderate and severe pain sensations (in accordance). The stimuli were given in a pseudo-random order twice, once before receiving the placebo pill (a sugar pill) and once after, maintaining the same order as before.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Sugar pill

SUMMARY:
Good clinical care relies on precise evaluation of patients' conditions. Chronic pain and other neurological and psychiatric diagnoses pose challenges because their assessment depends on subjective patient-reported outcome measures (PROs). The investigators have recently developed the Focused Analgesia Selection Task (FAST), a method that allows assessing pain reporting accuracy. Preliminary results suggest that those who more accurately report their pain show diminished placebo response. The underlying mechanisms for this observation cannot be explained by current theories. Therefore, the investigators have conducted a pilot study to further characterize this relation in healthy population.

DETAILED DESCRIPTION:
Instruments and procedures:

Instruments All stimuli were applied by a contact-heat Thermal Sen-sory Analyzer 2001 system (Medoc, Ramat-Yishai, Israel) with a 30 x 30mm Peltier surface stimulator, which was attached by Velcro straps to the volar surface of the forearm of the subjects' hand.

Familiarization session At the beginning of the experimental session, all subjects underwent short training in order to familiarize them with the device and with the sensations evoked by the painful stimulation, and to train them to report their perceived pain intensity using the numerical pain scale. The training included exposure to three short contact-heat stimuli (44, 46.5, and 48°C), each lasting for 7 seconds from the time that the stimulation intensity reached the destination temperature. The thermode was moved following each stimulus to a completely distinct, adjacent area of skin. Subjects were asked to report the numerical pain score (NPS), on a scale ranging from 0, denoting no pain, to 100, denoting the worst pain imaginable, induced by each stimulus.

Pain reporting accuracy assessment:

The subject's pain reporting accuracy skills was assessed by the FAST, which is based on recording a subject's pain reports in response to repeated administration of thermal noxious stimuli of various intensities. During the FAST procedure the thermode was attached to the ventral surface of the subject's non-dominant arm and the temperature was raised from a baseline of 32°C, peaked for 3 seconds at 1 of 7 designated temperatures (44°C, 45°C, 46°C, 47°C, 48°C, 49°C, and 50°C), and then decreased down to the baseline. Stimulus rate of rise and fall was kept constant at 8°C/seconds. Subjects were asked to rate the peak pain intensity of each stimulus verbally using the NPS. Each temperature was presented 7 times in a random block-ordered design (49 stimuli in total). Inter-stimulus intervals of 20 seconds allowed the subject sufficient time to rate the pain they perceived during each stimulus. The location of the thermode was adjusted every 10 stimuli to minimize sensitization and/or habituation effects. The duration of the FAST procedure is ~25 minutes.

Placebo assessment:

The placebo effect was assessed using tonic heat delivered at fixed temperature of either 44, 46.5, and 48°C. As was shown by previous studies, these temperatures evokes mild, moderate and severe pain sensations. During the stimuli, the thermode was attached to the volar surface of the forearm of the subjects' dominant hand. Baseline temperature was 32.0 °C, with an increasing temperature rate of 2°C/s and a return-to-baseline temperature rate of 8°C/s. Pain intensity ratings of heat stimuli were assessed verbally using NPS, at 2, 10 and 20 sec after the initiation of the stimulus.

Placebo procedure:

Each subject received clinical trial-type instructions before receiving the placebo so that the condition of the study would be similar to those encountered in typical drug trials. Subjects consented to participate in a study examining the analgesic effects of a well-known established pain relief medication. The subjects were told that they were about to receive a pain relief medication, which is commonly used in clinical practice. Possible adverse effects of the substance in question were then described, but it was indicated that the investigators did not typically observe significant adverse effects. Actual pharmacological agents were not administered.

Study design:

All experiments were conducted in the same setting, by the same investigator. The experiment was performed in a quiet room with an ambient temperature of 23°C. After the familiarization stage, the experiment begun with delivery of the FAST. After a 10 min break, subjects received the three tonic heat stimuli, each lasting 20 sec long, in a pseudo-random order with 60 sec break between each stimulus. Thereafter each subject was given a placebo pill. In order to evaluate placebo effect, the tonic heat stimuli were administered 20 minutes after placebo intake maintaining the same stimuli order.

The net placebo effect (Δ) was calculated as the difference between the mean NPS of the mild, moderate, and severe pain stimuli administrated before the placebo (Pre-placebo) minus the same after placebo (Post-placebo). The placebo effect in percent was calculated as the ratio of Post-placebo to Pre-placebo double 100. Positive values indicate efficient placebo effect.

The total duration of the experimental session was approximately 1 hours and 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* absence of acute or chronic pain disorders;
* no reports of psychiatric, cognitive and /or neurological disorders;
* no drugs including, analgesics or anti-anxiety medications on regular use (except for oral contraceptives).

Exclusion Criteria:

* pregnant or breast-feeding;
* unable to give informed consent, communicate and understand the purpose and the instructions of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-08-13 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Pain reporting accuracy | Fast procedure itself (49 heat stimuli, from 7 designated heat temperatures, given in a random block-order design) lasting approximately 20 minutes.
  Subjects will be asked to report their pain on numerical pain scale (NPS) ranging from 0, denoting "no pain", to 10, denoting "the worst pain imaginable".
Change in experimental pain perception due to placebo pill intake | Tonic stimuli before the placebo (Pre-placebo) until receiving the same stimuli 20 minutes after taking the placebo pill (Post-placebo).
  Subjects will be asked to report their pain on numerical pain scale (NPS) ranging from 0, denoting "no pain", to 10, denoting "the worst pain imaginable". The placebo effect (Δ) will be calculated as the difference between the mean NPS.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Haifa, The Clinical Pain Innovation Lab, Haifa, Israel